CLINICAL TRIAL: NCT04951505
Title: A Phase 1 Study to Evaluate the Safety and Intrapulmonary Pharmacokinetics of Cefepime and Taniborbactam in Healthy Subjects
Brief Title: Safety and Intrapulmonary Pharmacokinetics of Cefepime and Taniborbactam in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Venatorx Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VNRX-5133-107
Record Dates: First submitted 2021-06-28; First posted 2021-07-06 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- cefepime-taniborbactam (Experimental)
  Interventions: Drug: cefepime-taniborbactam

INTERVENTIONS:
Drug: cefepime-taniborbactam — IV infusion

SUMMARY:
This is a single-center, open-label study to assess the safety and intrapulmonary pharmacokinetics of cefepime and taniborbactam in healthy adult male and female subjects. Thirty subjects will receive a total of 6 doses of cefepime-taniborbactam (2 g cefepime/0.5g taniborbactam) administered intravenously every 8 hours. Following the sixth dose of cefepime-taniborbactam, subjects will be assigned to one of six bronchoscopy sampling times.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults 18-55 years
2. Males or non-pregnant, non-lactating females
3. Body mass index (BMI): ≥18 kg/m2 and ≤32.0 kg/m2, weight >50.0 kg.
4. Must have negative alcohol, drug, or tobacco use/test and no use of alcohol, caffeine during the study

Exclusion Criteria:

1. History or presence of current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, autoimmune, hematologic, neoplastic, or neurological disorders
2. History of drug allergy or hypersensitivity to penicillin, cephalosporin, or beta-lactam antibacterial drug
3. Recent history of known or suspected Clostridioides difficile infection
4. Abnormal ECG or history of clinically significant abnormal rhythm disorder
5. Abnormal lab tests

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
ELF Cmax | 0-8 hours after 6th dose
  Maximum concentrations of cefepime and taniborbactam, determined directly from individual concentration-time data, in epithelial lining fluid (ELF)

SECONDARY OUTCOMES:
Number of subjects with adverse events | Day 1 - Day 8

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonary Associates PA, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Rodvold KA, Gotfried MH, Sabato P, Henkel T, McGovern PC. Plasma and intrapulmonary pharmacokinetics of cefepime and taniborbactam in healthy adult participants. Antimicrob Agents Chemother. 2025 Jul 2;69(7):e0049325. doi: 10.1128/aac.00493-25. Epub 2025 Jun 6. PMID 40476839